CLINICAL TRIAL: NCT04817163
Title: Implementation of a Stepped Care Cognitive-Behavioral Therapy for Insomnia in Routine Cancer Care
Brief Title: Implementation of CBT-I in Cancer Clinics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Josée Savard, Researcher, CHU de Quebec-Universite Laval
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IC118713
Record Dates: First submitted 2021-03-18; First posted 2021-03-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Insomnia
Keywords: Insomnia; Cancer; Cognitive-behavioral therapy; Stepped care model; Self-administered treatment; Web-based intervention; Implementation; Cost-effectiveness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Neoplasms

STUDY DESIGN:
Intervention Model Description: The stepped care CBT-I (active intervention) is being implemented sequentially in the four participating hospitals over a number of equally spaced time periods of 4 months (wedges), for a total of 5 time points, over a period of 20 months.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stepped care CBT-I (Experimental)
  Interventions: Behavioral: Web-based cognitive-behavioral therapy for insomnia (CBT-I); Behavioral: Professionally-administered booster face-to-face CBT-I sessions

INTERVENTIONS:
Behavioral: Web-based cognitive-behavioral therapy for insomnia (CBT-I) — Each week, the patients first have to read written information on the website (www.insomnet.ca), and then watch a video capsule (duration between 5 and 20 min each). Patients complete their daily sleep diary electronically on the website and the content is interactive. It includes the sending of automated emails to remind participants to complete the treatment tasks and encourage adherence, provision of tailored feedback (e.g., texts, charts) based on the information that they provide in their sleep diary, as well as quizzes with automated correction to reinforce patients' understanding of the content.
  Other Names: Self-administered
Behavioral: Professionally-administered booster face-to-face CBT-I sessions — Patients who obtain an ISI score of 8 and more after completing the web-based CBT-I are "stepped up" and offered to receive up to three 50-min booster sessions of CBT-I offered individually by a psychologist (if needed). Remitted patients (good sleepers; ISI score lower than 8) will receive no further treatment.

SUMMARY:
Insomnia affects 30-60% of cancer patients, thus making it one of the most common disturbances in this population. When untreated, which is the rule rather than the exception, insomnia often becomes chronic. Chronic insomnia is associated with numerous negative consequences (e.g., increased risk for psychological disorders, health care costs). A large body of evidence supports the efficacy of cognitive-behavioral therapy for insomnia (CBT-I) in cancer patients, but CBT-I is still not offered routinely in cancer clinics. Self-administered CBT-I (e.g., video-based intervention) has been developed to increase patients' access to this treatment. However, results of clinical trials have suggested that these minimal treatments would be better used as a first step of a stepped care model. In stepped care, patients receive only the level of intervention they need. Generally, the entry level is a minimal, less costly, intervention (e.g., self-help intervention) followed by a more intensive form of treatment if needed (if the patient is still symptomatic). The investigators have recently assessed the efficacy of a stepped care model to administer CBT-I in cancer patients, which includes a web-based CBT-I (called Insomnet) followed by up to 3 sessions with a psychotherapist if the patient is still symptomatic. Results of this study suggest that this model of care is non-inferior to a standard face-to-face treatment (Savard, Ivers, et al., in revision), while being more cost-effective. A stepped care CBT-I could therefore be offered in routine cancer care clinics.

This project will assess the feasibility and effectiveness of implementing a stepped care CBT-I in real-world cancer clinics, using a non-randomized stepped wedge design to compare the effects of our program (active phase) with a passive phase. The program is called Insomnia in Patients with Cancer - Personalized Treatment (IMPACT). The stepped care CBT-I (active intervention) is being implemented sequentially in the four participating hospitals over a number of equally spaced time periods of 4 months (wedges), for a total of 5 time points, over a period of 20 months.

ELIGIBILITY:
Inclusion Criteria:

* have received a diagnosis of non-metastatic cancer (any type)
* to be aged 18 years and older
* to be readily able to read and understand French or English
* having the minimum cognitive abilities to read, understand and memorize information
* having access to Internet

Exclusion Criteria:

* having a psychological comorbidity needing clinical attention (e.g., major depressive disorder)
* having severe cognitive impairments (e.g., diagnosis of Parkinson's disease, dementia)
* having insomnia due to a temporary condition (e.g., acute pain, short-term medication side effects, environmental factors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Implementation (organizational) measures | Passive phase (4 months) vs. active phase (20 months), through study completion, an average of 24 months
  Referral, enrolment and completion rates to the stepped care CBT-I in each clinical setting.
1) Change in Insomnia Severity Index Scores | Pre-treatment and post-treatment (6-8 weeks later)
  Change in Insomnia Severity Index Scores from pre- to post-intervention. The ISI is a 7-item questionnaire designed to evaluate insomnia severity. A score greater than or equal to 8 indicates the presence of insomnia symptoms.
2) Change in sleep efficiency (SE) | Pre-treatment and post-treatment (6-8 weeks later)
  Change in daily sleep diary parameters from pre- to post-intervention: Change in sleep efficiency (SE) index (%) = Total sleep time/total time spent in bed X 100.
3) Change in sleep onset latency (SOL) | Pre-treatment and post-treatment (6-8 weeks later)
  Change in daily sleep diary parameters from pre- to post-intervention: Change in sleep onset latency (SOL) = Time to sleep after lights out.
4) Change in wake after sleep onset (WASO) | Pre-treatment and post-treatment (6-8 weeks later)
  Change in daily sleep diary parameters from pre- to post-intervention: Change in wake after sleep onset (WASO) = Summation of nocturnal awakenings.
5) Change in total wake time (TWT) | Pre-treatment and post-treatment (6-8 weeks later)
  Change in daily sleep diary parameters from pre- to post-intervention: Change in total wake time (TWT) = Summation of SOL, WASO, and early morning awakening.
6) Change in total sleep time (TST) | Pre-treatment and post-treatment (6-8 weeks later)
  Change in daily sleep diary parameters from pre- to post-intervention: Change in total sleep time (TST) = Time in bed minus total wake time.
7) Hospital Anxiety and Depression Scale (HADS) | Pre-treatment and post-treatment (6-8 weeks later)
  Change scores from pre to post-intervention: Hospital Anxiety and Depression Scale (HADS): A 14-item questionnaire comprising 7 items assessing depression and 7 items assessing anxiety. Scores obtained for each subscale range from 0 to 21.
8) Fatigue Symptom Inventory (FSI) | Pre-treatment and post-treatment (6-8 weeks later)
  Change scores from pre to post-intervention: Fatigue Symptom Inventory (FSI): A 14-item questionnaire measuring perceived fatigue. Each item is rated on an 11-point Likert scale, ranging from 0 to 10. A higher score indicates a higher level of fatigue or interference or a longer duration of fatigue.
9) The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Pre-treatment and post-treatment (6-8 weeks later)
  Change scores from pre to post-intervention: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30): A 30-item questionnaire. Scores are transformed to give a score ranging from 0 to 100.
10) Satisfaction with Life Scale (SWLS) | Pre-treatment and post-treatment (6-8 weeks later)
  Change scores from pre to post-intervention: Satisfaction with Life Scale (SWLS): A 5-item questionnaire (Likert scale from 1 to 7) designed to measure global cognitive judgments of satisfaction with one's life.
1) Psychologists' adherence to the protocol | Throughout the active phase, up to 20 months
  Psychologists' self-assessed adherence to the CBT-I protocol (%)
2) Psychologists' perceived self-efficiency | Throughout the active phase, up to 20 months
  Psychologists' perceived self-efficiency in using CBT-I protocol (%)

SECONDARY OUTCOMES:
1) Demographic characteristics | Pre-treatment and post-treatment (6-8 weeks later) for patient; Through study completion (an average of 24 months) for clinicians
  Clinicians and patients' demographics (e.g., age, sex)
2) Evidence-Based Practice Attitudes Scale (EBPAS) | Through study completion, an average of 24 months
  Administrators' and clinicians' attitude towards empirically-based treatments (Evidence-Based Practice Attitudes Scale (EBPAS; 15 items)): Scores obtained range from 0 to 60.
3) Workplace Stress Scale (WSS) | Through study completion, an average of 24 months
  Stress at work (Workplace Stress Scale (WSS; 8 items)): Scores obtained range from 8 to 40.
4) Organizational Readiness for Implementing Change (ORIC) | Through study completion, an average of 24 months
  Attitude towards change (Organizational Readiness for Implementing Change (ORIC; 12 items)): Participants rated the hospital's readiness for implementation on 12 items using a 5-point ordinal scale that ranged from "disagree" (1) to "agree" (5).
5) Clinicians expertise | Through study completion, an average of 24 months
  Clinicians' CBT expertise (number of years of experience with CBT)
6) Internet Evaluation and Utility Questionnaire (IEUQ) | Pre-treatment and post-treatment (6-8 weeks later)
  Patients' familiarity with the Internet (Internet Evaluation and Utility Questionnaire (IEUQ; 15 items)): Patients respond to the questions on a 5-point likert scale from "not at all" (0) to "very" (4), with 2 open-ended items asking patients to identify "most helpful" and "least helpful" parts of the web program.
7) Brief Health Literacy Screening Tool (BRIEF) | Pre-treatment and post-treatment (6-8 weeks later)
  Health literacy (Brief Health Literacy Screening Tool (BRIEF; 4 items)): Each item ranges from 1 to 5 and total scores range from 4 to 20.
Possible moderating treatment effect | Pre-treatment (at recruitment)
  Possible moderating treatment effect by some of the participants' characteristics (e.g., age, sex, cancer site).

CONTACTS AND LOCATIONS:
Overall Officials: Josée Savard, Ph.D., Principal Investigator — Centre de recherche du CHU de Québec-Université Laval
Locations (1):
- Centre de recherche de L'Hôtel-Dieu de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No